CLINICAL TRIAL: NCT04157764
Title: The Impact of Telemonitoring on Compliance and Outcomes of Patients Undergoing Automated Peritoneal Dialysis With SHARESOURCE
Brief Title: Improve Compliance in Automated Peritoneal Dialysis Machine With SHARESOURCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: E-DA Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMRP108057
Record Dates: First submitted 2019-10-14; First posted 2019-11-08 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Compliance, Patient
Keywords: Telehealth; automated peritoneal dialysis
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Intervention Model Description: use automated peritoneal dialysis machine without SHARESOURCE for 12 weeks, then use automated peritoneal dialysis machine with SHARESOURCE for 12 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- APD (Experimental)
  Interventions: Device: HomeChoice Claria APD machine with SHARESOURCE

INTERVENTIONS:
Device: HomeChoice Claria APD machine with SHARESOURCE — HomeChoice Claria APD machine with SHARESOURCE software. SHARESOURCE is a software can telemonitor patients' compliance

SUMMARY:
This study is to investigate the non-compliance rate of patients undergoing automated peritoneal dialysis by using automated peritoneal dialysis with SHARESOURCE software, and to evaluate if telemonitoring can improve peritoneal dialysis compliance and outcomes in the observation period.

DETAILED DESCRIPTION:
The non-compliance of patients receiving automated peritoneal dialysis (APD) is around 10-20%, and was believed to be under-estimated. Recently, a two-way telehealth system, SHARESOURCE software, provide practitioners real-time monitoring and recording of the therapy of APD.

By using this APD with SHARESOURCE software, we want to investigate the non-compliance rate of patients undergoing automated peritoneal dialysis, want to see if it can improve peritoneal dialysis compliance and outcomes in the observation period.

ELIGIBILITY:
Inclusion Criteria:

* stable received peritoneal dialysis for over 1 year. Use automated peritoneal dialysis machine regularly by him/herself.

Exclusion Criteria:

* Acute hospitalization events due to acute coronary syndrome, stroke, heart failure, liver cirrhosis, systemic infection in 1 month.
* Life expectancy <1 year
* Peritoneal dialysis prescriptions will be scheduled or expected to change in 3 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2021-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Change of baseline patients' non-compliance rate at 3 months | baseline(between week 0 and 12) and 3 months(week 12 and week 24)
  Non compliance rate was calculated by the days of non-compliance divided by days of APD therapy

SECONDARY OUTCOMES:
Change of baseline peritoneal dialysis adequacy at 3 and 6 months | baseline, week 12 and week 24
  Dialysis adequacy is to see if dialysis is enough
Change of baseline uremic toxin level at 3 and 6 months | baseline, week 12 and week 24
  concentration of uremic toxins(ex: indoxyl sulfate, and p-cresyl sulfate)
change of body composition analysis | baseline, week 12 and week 24
  body composition exam (Body Composition Monitor, Fresenius Medical Care, Bad Homburg, Germany) will be done
peritonitis rate (patient-month) | follow up to week 60
  calculate the number of peritonitis rate
Hospitalization rate | follow up to week 60
  calculate the number of hospitalization rate
Change of telephone contact frequency | baseline(between week 0 and 12) and 3 months(week 12 and week 24)
  the telephone contact frequency (from patient to nurse) for peritoneal dialysis-related problems will be collected

REFERENCES:
- [Background] Saran R, Robinson B, Abbott KC, Agodoa LYC, Bragg-Gresham J, Balkrishnan R, Bhave N, Dietrich X, Ding Z, Eggers PW, Gaipov A, Gillen D, Gipson D, Gu H, Guro P, Haggerty D, Han Y, He K, Herman W, Heung M, Hirth RA, Hsiung JT, Hutton D, Inoue A, Jacobsen SJ, Jin Y, Kalantar-Zadeh K, Kapke A, Kleine CE, Kovesdy CP, Krueter W, Kurtz V, Li Y, Liu S, Marroquin MV, McCullough K, Molnar MZ, Modi Z, Montez-Rath M, Moradi H, Morgenstern H, Mukhopadhyay P, Nallamothu B, Nguyen DV, Norris KC, O'Hare AM, Obi Y, Park C, Pearson J, Pisoni R, Potukuchi PK, Repeck K, Rhee CM, Schaubel DE, Schrager J, Selewski DT, Shamraj R, Shaw SF, Shi JM, Shieu M, Sim JJ, Soohoo M, Steffick D, Streja E, Sumida K, Kurella Tamura M, Tilea A, Turf M, Wang D, Weng W, Woodside KJ, Wyncott A, Xiang J, Xin X, Yin M, You AS, Zhang X, Zhou H, Shahinian V. US Renal Data System 2018 Annual Data Report: Epidemiology of Kidney Disease in the United States. Am J Kidney Dis. 2019 Mar;73(3 Suppl 1):A7-A8. doi: 10.1053/j.ajkd.2019.01.001. Epub 2019 Feb 21. No abstract available. PMID 30798791
- [Background] Bernardini J, Piraino B. Compliance in CAPD and CCPD patients as measured by supply inventories during home visits. Am J Kidney Dis. 1998 Jan;31(1):101-7. doi: 10.1053/ajkd.1998.v31.pm9428459.
- [Background] The USRDS Dialysis Morbidity and Mortality Study: Wave 2. United States Renal Data System. Am J Kidney Dis. 1997 Aug;30(2 Suppl 1):S67-85. No abstract available. PMID 9259694
- [Background] Milan Manani S, Crepaldi C, Giuliani A, Virzi GM, Garzotto F, Riello C, de Cal M, Rosner MH, Ronco C. Remote Monitoring of Automated Peritoneal Dialysis Improves Personalization of Dialytic Prescription and Patient's Independence. Blood Purif. 2018;46(2):111-117. doi: 10.1159/000487703. Epub 2018 Apr 25. PMID 29694954
- [Background] Uchiyama K, Washida N, Yube N, Kasai T, Shinozuka K, Morimoto K, Hishikawa A, Inoue H, Urai H, Hagiwara A, Fujii K, Wakino S, Deenitchina S, Itoh H. The impact of a remote monitoring system of healthcare resource consumption in patients on automated peritoneal dialysis (APD): A simulation study . Clin Nephrol. 2018 Nov;90(5):334-340. doi: 10.5414/CN109471. PMID 30106369